CLINICAL TRIAL: NCT03586908
Title: An Open Label, Multiple-dose, Phase 1 Clinical Trial to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of PHP-201 Topical Eye Drop in Korean and Japanese Healthy Subjects
Brief Title: PK/PD, Safety and Tolerability of PHP-201 Topical Eye Drop in Korean and Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pH Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHP-201-S102
Record Dates: First submitted 2018-04-19; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — sovesudil; Ophthalmic Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PHP-201 0.5% (Experimental): PHP-201 0.5%, ophthalmic solution, topical eye drop, OU
  Interventions: Drug: PHP-201 0.5% ophthalmic solution (topical eye drop)

INTERVENTIONS:
Drug: PHP-201 0.5% ophthalmic solution (topical eye drop) — D1, D7: PHP-201 0.5% topical eye drop OU QD(AM), D2~D6: PHP-201 0.5% topical eye drop OU TID
  Other Names: PHP-201 5mg/ml

SUMMARY:
An open label, multiple-dose, phase 1 clinical trial to evaluate pharmacokinetics, pharmacodynamics, safety and tolerability of PHP-201 topical eye drop in Korean and Japanese healthy subjects

DETAILED DESCRIPTION:
Primary: The evaluation of pharmacokinetic properties of repeating PHP-201 topical eye drop Secondary: The evaluation of pharmacodynamic, safety and tolerability of repeating PHP-201 topical eye drop

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed about the purpose of the study
2. BMI of 18.0 kg/m² or more and 27.0 kg/m² or less who are between 19 and 50 years of age
3. No congenital or chronic disease and no medically symptomatic findings

Exclusion Criteria:

1. Clinically significant disease history or disease history that may affect the absorption, distribution, metabolism and excretion of the drug, or ophthalmic corneal surgery
2. had BCVA worse than logMAR 0.2(20/30snellen) or IOP < 10mmHg or >21mmHg in either eye
3. Abnormalities of clinical examination (SBP, DBP, pulse rate, AST, ALT, Total bilirubin, eGFR and Serum test, ECG)
4. Allergy, drug hypersensitivity and substance abuse
5. Forbidden drug and diet
6. Blood donation and transfusion

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 1week
  Cmax of PHP-201 & Metabolite
Time to Cmax[Tmax] | 1week
  Tmax of PHP-201 & Metabolite

SECONDARY OUTCOMES:
Mean Change of Intraocular pressure(IOP) | 1week
  Mean Change from baseline IOP after 1week

CONTACTS AND LOCATIONS:
Overall Officials: Soojin Kim, Study Director — pH Pharma
Locations (1):
- Inje University Busan Baek Hospital, Busan, Busanjin-gu, South Korea

IPD SHARING:
Plan to Share IPD: No